CLINICAL TRIAL: NCT00949195
Title: Pulmonary Arterial Pressure Response During Exercise in COPD and Healthy Subjects
Brief Title: Pulmonary Arterial Pressure Response During Exercise
Acronym: PAPCOPDHS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Attila Somfay, MD, PhD; Department Leader, Department of Pulmonology, Szeged University
Other Study IDs: SZTE PULM-PAHP; ISRCTN11034505
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2009-10

CONDITIONS: COPD Patients; Healthy Subjects; Semi-supine Echo (SSE); Flow-mediated Vasodilatation (FMD); High Sensitive C-reactive Protein (hsCRP)
Keywords: COPD; healthy patients; PAP; CPX; SSE; hsCRP; FMD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ventilation; C-Reactive Protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood sample is taken to analyse the systemic inflammatory marker (hsCRP) level from serum. We measure the samples and than we don't store it.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- COPD patients: COPD patients with severe obstruction performed the tests.
  Interventions: Other: Measure pulmonary artery pressure change during exercise; Other: Pulmonary pressure response during exercise
- Healthy subjects: Age-matched healthy subjects performed the same test also.
  Interventions: Other: Measure pulmonary artery pressure change during exercise; Other: Pulmonary pressure response during exercise

INTERVENTIONS:
Other: Measure pulmonary artery pressure change during exercise — Semi-supine echocardiography test
  Other Names: lung function, CPX, HsCRP
Other: Pulmonary pressure response during exercise — Semi-supine echocardiography test
  Other Names: Complete lung function, CPX, HsCRP

SUMMARY:
Background:

The extent of increase in systolic pulmonary arterial pressure (PAPs) during exercise in patients with COPD is unpredictable from lung function data. The non-invasive assessment of pulmonary hemodynamics during exercise and flow-mediated vasodilatation measurement may give useful data in the rehabilitation of COPD patients.

Methods:

Patients with stable, severe COPD and healthy, age-matched subjects (H) perform semi supine echocardiography with PAPs measurement. COPD patients perform ramp protocol with gas exchange detection. Serum hsCRP level is also determined in COPD patients. Endothel dysfunction is detected by flow mediated vasodilation measurement after arm strangulation with Doppler ultrasonography.

Primary endpoint:

The degree of pulmonary artery systolic pressure change during exercise?

Secondary endpoint:

1. The degree of right ventricular function change during exercise?
2. Is endothel dysfunction manifested with pulmonary artery pressure rise?
3. What is the correlation between the systemic inflammatory marker hsCRP and the degree of pulmonary artery pressure rise?

DETAILED DESCRIPTION:
Background: The extent of increase in systolic pulmonary arterial pressure (PAPs) during exercise in patients with COPD is unpredictable from lung function data. The non-invasive assessment of pulmonary hemodynamics during exercise by semi-supine echocardiography and flow-mediated vasodilatation measurement may give useful data in the rehabilitation of COPD patients.

Methods: Patients with stable, severe COPD and healthy, age-matched subjects (H) perform semi supine echocardiography with PAPs measurement. COPD patients perform ramp protocol with gas exchange detection. Serum hsCRP level is also determined in COPD patients. All of the subjects perform complete lung function with body pletysmography and diffusion capacity measurement. Endothel dysfunction is detected by flow mediated vasodilation measurement after arm strangulation with Doppler ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (age between 45 and 70)
* with moderate to severe obstruction (FEV1<60%pred) and
* healthy subjects (age between 45 and 70, (FEV1>80%pred, FEV1/FVC>70%

Exclusion Criteria:

* Not in the age range
* Different FEV1 value
* Severe comorbidities

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients (age between 45 and 70) with moderate to severe obstruction (FEV1<60%) and healthy subjects (age between 45 and 70)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-12; Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The degree of pulmonary artery pressure change during exercise? | 2 months

SECONDARY OUTCOMES:
Right ventricular function change? Correlation between systemic inflammation (hsCRP) and pulmonary artery pressure change? Endothelial dysfunction? | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Attila Somfay, MD, PhD, Principal Investigator — Department of Pulmonology, Szeged University
Locations (1):
- Department of Pulmonology, Szeged University, Deszk, Csongrád megye, Hungary

REFERENCES:
- [Derived] Varga J, Palinkas A, Lajko I, Horvath I, Boda K, Somfay A. Pulmonary Arterial Pressure Response During Exercise in COPD: A Correlation with C-Reactive Protein (hsCRP). Open Respir Med J. 2016 Jan 29;10:1-11. doi: 10.2174/1874306401610010001. eCollection 2016. PMID 27019674